CLINICAL TRIAL: NCT05516355
Title: Psychological and Neurobiological Impact of a Retreat Based on Mindfulness and Compassion for Stress Reduction.
Acronym: Retreat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Carmelo Vázquez, Full Professor of Psychopathology, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ESCORIAL RETREAT 2022
Record Dates: First submitted 2022-08-21; First posted 2022-08-25 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Mindfulness; Compassion; Psychophysiologic Reaction; Psychological Distress; Emotion Regulation; Stress
Keywords: MBSR; CCT; Mindfulness; Compassion; Epigenetics; Stress
MeSH Terms: conditions — Emotional Regulation | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: MBSR and CCT instructors will be blind to the study hypotheses. Investigators collecting, analyzing data and assessing outcomes will be blind to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (MBSR + CCT) (Experimental): Group 1 will begin the retreat with a 3-day MBSR intervention. On day 4 of the retreat, they will crossover and begin a 3-day CCT intervention.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction; Behavioral: Compassion Cultivation Training
- Group 2 (CCT + MBSR) (Experimental): Group 2 will begin the retreat with a 3-day CCT intervention. On day 4 of the retreat, they will crossover and begin a 3-day MBSR intervention.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction; Behavioral: Compassion Cultivation Training

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The MBSR is an 8-week standardized program (Kabat-Zinn,1990).
  During the retreat, participants will receive intensive training during 3 days (from 4:00pm to 9pm the first day and from 7 am to 10 pm including breaks, the second and third days), including focused attention on the breath, open monitoring of awareness in body-scanning, prosocial meditation (i.e. loving kindness and compassion) and gentle yoga. Training is delivered by certified instructors by the University of Massachusetts Centre for Mindfulness (https://www.umassmed.edu/cfm/).
  Other Names: MBSR
Behavioral: Compassion Cultivation Training — The CCT is an 8-week standardized program (Jinpa, 2010; Jazaieri et al. 2013, 2014) consisting of daily formal and informal practices.
  Training will be conducted during 3 days of the retreat (same schedule as the MBSR training). The CCT consists of six sequential steps: 1) Settling the mind and learn how to focus it; 2) Loving kindness and compassion for a loved one practice; 3) Loving kindness and compassion for oneself practice; 4) compassion toward others, embracing shared common humanity and developing appreciation of others; 5) compassion toward others including all beings; and 6) active compassion practices (Tonglen) which involve explicit evocation of the altruistic wish to do something about others' suffering. CCT program is delivered by certified instructors by the University of Stanford Centre for Compassion and Altruism Research and Education (http://ccare.stanford.edu/).
  Other Names: CCT

SUMMARY:
The study is aimed at comparing the differential effects of two widely used standardized meditation programs: Mindfulness-Based Stress Reduction (MBSR) and Compassion Cultivation Training (CCT) delivered in a retreat format with a cross-over design in a general population sample of healthy adults.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effects of two mindfulness-based intensive interventions: Mindfulness-Based Stress Reduction (MBSR) training or Compassion Cultivation Training (CCT), on psychological, physiological and epigenetic changes in a population of health volunteer adults. During a 7-day retreat participants will be randomised to two study arms: group 1 and 2, beginning either with a 3-day MBSR training or a 3-day CCT training. On the 4th day they will cross-over to the opposite intervention.

To address this goal, the effects will be measured by self-report questionnaires belonging to different domains (mindfulness, compassion, well-being, psychological distress, and psychological functioning), psychophysiological measures (EEG resting state, Diurnal cortisol slope, EKG and respiration patterns), epigenetic changes (DNA methylation biomarkers) and an objective stress task (Arithmetic Stress Test). Psychobiological outcome measures will be collected from both groups on day 1 (pre-intervention), on day 4 (post intervention and before beginning of the second intervention). The third assessment will be conducted on day 7 for both groups (post-second intervention). A 6-month follow-up assessment will be carried in both groups only for psychological questionnaires.

Data analysis will include change scores in psychological outcome measures as well as DNA methylation (by EPIC arrays) and gene expression (RNA-seq) measures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants.

Exclusion Criteria:

* Current or past self-reported diagnosable serious or disabling mental disorder (in particular, PTSD, major depression, psychotic disorders, and/or Use of alcohol or drugs disorders).
* Presenting current health conditions that might affect the immune system (i.e. autoimmune disease, chronic severe infections, HIV, cancer) or past history of the same (less than 5 years from total recovery).
* Presenting current habits that might affect the immune system (i.e. smoking, alcoholism, substance abuse).
* Being under medical treatment that might affect the immune system response and inflammatory processes (i.e. corticoids).
* Travelling from a different time zone/long-travel times that might affect the immune system.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Epigenetic changes | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  Blood samples: 20 ml collected in the standard tubes used in clinical haematology that contain EDTA as an anticoagulant. From this biological material, DNA and RNA will be extracted according to the standard molecular biology procedures, in order to subsequently measure DNA methylation (by EPIC arrays) and gene expression (RNA-seq), respectively.
Change in Psychological distress | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  Depression Anxiety Stress Scales (DASS-21), (Lovibond and Lovibond, 1995). The DASS-21 is a 21-item scale containing 3 subscales (Anxiety, Depression and Stress), with 7 items for each subscale. Participants are asked to rate each item using 4-point Likert scale (0=Not applicable to me; 3=Very applicable to me). Higher scores correspond to higher levels of severity of anxiety, stress, and depression.
Change in Stress Reactivity | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  Mathematical Stress Test: a standardized laboratory stress induction procedure (Kirshbaum et al., 1992). Individuals are asked to repeatedly subtract a given 2-digit number from a 4-digit number. Time is limited to 3 minutes and participants are told that this is a mental speed task and their performance will be evaluated. Stress levels will be evaluated with an affective adjective checklist (PANAS scales).
Change in Resting State Activity | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  EEG resting state (alternating open and closed eyes). EEG resting state will be recorded with four 64-channel EEG devices with laptop and eego EEG recording software. The sampling rate will be 1000 Hz and the reference to be used will be 7Z of the equidistant layout.
  The interventions will significantly change the EEG spectral profile of the resting state brain activity. We expect changes in the balance between Alpha (8-14 Hz) and Theta (4-8 Hz) frequency bands.
Change in Cortisol activity | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program
  Cortisol samples 1.5 - 2.0 ml will be collected in Salivette® cortisol saliva sample collection tubes (Sarstedt, Germany) that contain sterile cotton plugs for sample absorption. From this biological material, levels of the principal stress corticosteroid, the hormone cortisol, will be assessed in order to subsequently measure the Diurnal Cortisol Slope and cortisol levels at awakening and bedtime.
  Using saliva collection tubes, levels of the principal stress corticosteroid, the hormone cortisol, will be assessed in order to subsequently measure the Diurnal Cortisol Slope and cortisol levels at awakening and bedtime at three different moments of the retreat.
Change in Emotion regulation in retrieving autobiographical negative memories | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  A 10-min guided test to retrieve one personally painful memory. Affect changes will be asssed before and after the task by using a checklist of affective adjectives (PANAS).

SECONDARY OUTCOMES:
Change in Mindfulness State | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  State Mindfulness Scale (SMS) - (Tanay y Bernstein, 2013). The SMS has 21 items with a response scale from 1 (not at all) to 5 (very well) to indicate how well the statements describe their current mindfulness state. Higher scores represent higher states of current mindfulness.
Change in Mindfulness - Adverse Effects | Mid-intervention (T2: Day 4 in the 7-day program), post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  Meditation-Related Adverse Effects Scale - Mindfulness-Based Program (MRAESMBP) -Britton et al. (2018). This is an 11-item scale measuring the frequency of challenging or distressful experiences during meditation practice.
Change in Compassion - State self-compassion | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  State Self-compassion Scale (SSCS), (Neff et al., 2021). It is a 6-item scale measuring compassion towards oneself using a 5-'point scale (1=Not at all true for me; 5= Very true for me). HIgher scores indicate higher levels of self-compassion.
Change in Compassion - Fear of Compassion | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  We will use the Fear of Expressing Compassion towards yourself subscale from the Fear of Compassion Scale (Gilbert et al. (2011). This is a 15-item scale to assess individuals' difficulties to feel or express self-compassion. We by using a 5-point Likert scale (0=Don't agree at all; 4=Completely agree). Higher scores indicate higher levels of fear of compassion towards oneself.
Change in current mood | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  A scale measuring current general positive and negative mood (PANAS). It includes 20 adjectives (10 positive, 10 negative) to assess current mood in a scale from 1 (Not all) to 5 (Extremely). Higher scores represent higher positive or negative mood states. We will use the sum of positive items and negative items to provide two separate overall scores.
Change in Psychological well-being - Satisfaction with life | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  Satisfaction With Life Scale (SWLS), (Diener et al., 1985). This is a 5-item scale assessing satisfaction with life. Higher scores indicate higher levels of satisfaction with life.
Change in Somatic Symptoms | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  Patient Health Questionnaire (PHQ-15), (Kroenke et al., 2002). The PHQ-15 comprises 15 somatic symptoms from the PHQ, each symptom scored from 0 ("not bothered at all") to 2 ("bothered a lot"). A sum score will be used to analyze somatic symptoms.
Change in Emotion Regulation | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  State Difficulties in Emotion Regulation (S-DERS-21), (Lavender et al., 2017). This is a 21-item scale in which participants rate their difficulties to regulate their mood in a 5-point Likert scale (1=Not alll; 5=Completely). Higher scores indicate more difficulties in emotion regulation.
Change in Anxiety state and trait | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  State-Trait Anxiety Inventory (STAI-20), (Spielberger et al., 1983)
Change in Sleep difficulties | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  DSM-5 sleep difficulties (APA, 2013). This is the single item included in the Self-rated level 1 Cross-Cutting Symptom Measure (DSM-5, APA 2013). It measures quality of sleep using a 5-point scale (0=Very good; 4= Very bad).
Program satisfaction | Mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  Client Satisfaction Questionnaire (CSQ-8)- Atkinson and Zwicq (1982). It measures satisfaction with the course of psychological interventions. Participants must rate their satisfaction on 8 items in 4-point scale. Higher scores indicate higher satisfaction with the program.
Daily assessments of psychological functioning | Daily, at the end of the day, during the 7-day retreat
  Experience Sampling Methods on measures of: mindfulness, mind wandering, compassion to others, self-compassion, wellbeing, richness of life, and utility of the contents of the program that day. These are 'ad hoc' single items, taken from well-validated measures, to have a quick daily assessment of psychological functioning. Each item is assessed in a 5-point Likert scale (0=Never; 4= Always).
Change in Affect | Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program), and 3-month follow-up (T4)
  Hedonic and Arousal Affect Scale (HAAS), (Roca et al., 2021). This is a 12-item scale measuring affective states by including adjectives low or high in arousal and positive or negative in valence. Participants are asked to rate their affective experiences in a 5-point Likert scale (0=Not at all; 4= Absolutely).

OTHER OUTCOMES:
EKG activity | ime Frame: Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  Measurement of cardiac activity during EEG sessions. EKG will be used in the preprocessing procedure to insulate electrophysiological artifacts due to heart activity. In addition, the heart signals will be assessed to obtain heart variability and heart rate indicators.
Respiratory patterns | ime Frame: Pre-intervention (T1: Day 1 in the 7-day program), mid-intervention (T2: Day 4 in the 7-day program), and post-intervention (T3: Day 7 in the 7-day program)
  Measurement of respiratory activity during EEG sessions. Respiratory signals will be employed in an specific analysis where the EEG data will be split in two blocks (inhalation and exhalation).

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Vazquez, Ph.D., Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid - Faculty of Psychology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez-Lopez MJ, Conklin QA, Cosin-Tomas M, Shields GS, King BG, Zanesco AP, Kaliman P, Saron CD. Changes in the expression of inflammatory and epigenetic-modulatory genes after an intensive meditation retreat. Compr Psychoneuroendocrinol. 2022 Jun 23;11:100152. doi: 10.1016/j.cpnec.2022.100152. eCollection 2022 Aug. PMID 35818436
- [Background] Bishop, S. R., Lau, M., Shapiro, S., Carlson, L., Anderson, N. D., Carmody, J., Segal, Z. v., Abbey, S., Speca, M., Velting, D., & Devins, G. (2004). Mindfulness: A proposed operational definition. Clinical Psychology: Science and Practice, 11(3), 230-241. https://doi.org/10.1093/clipsy/bph077
- [Background] Chambers, R., Lo, B. C. Y., & Allen, N. B. (2008). The impact of intensive mindfulness training on attentional control, cognitive style, and affect. Cognitive therapy and research, 32(3), 303-322. https://doi.org/10.1007/s10608-007-9119-0
- [Background] Chiesa A, Calati R, Serretti A. Does mindfulness training improve cognitive abilities? A systematic review of neuropsychological findings. Clin Psychol Rev. 2011 Apr;31(3):449-64. doi: 10.1016/j.cpr.2010.11.003. Epub 2010 Dec 1. PMID 21183265
- [Background] Cohen, J. N., Jensen, D., Stange, J. P., Neuburger, M., & Heimberg, R. G. (2017). The immediate and long-term effects of an intensive meditation retreat. Mindfulness, 8(4), 1064-1077.
- [Background] Davidson RJ, Kaszniak AW. Conceptual and methodological issues in research on mindfulness and meditation. Am Psychol. 2015 Oct;70(7):581-92. doi: 10.1037/a0039512. PMID 26436310
- [Background] Fransquet PD, Wrigglesworth J, Woods RL, Ernst ME, Ryan J. The epigenetic clock as a predictor of disease and mortality risk: a systematic review and meta-analysis. Clin Epigenetics. 2019 Apr 11;11(1):62. doi: 10.1186/s13148-019-0656-7. PMID 30975202
- [Background] Galante J, Friedrich C, Dawson AF, Modrego-Alarcon M, Gebbing P, Delgado-Suarez I, Gupta R, Dean L, Dalgleish T, White IR, Jones PB. Mindfulness-based programmes for mental health promotion in adults in nonclinical settings: A systematic review and meta-analysis of randomised controlled trials. PLoS Med. 2021 Jan 11;18(1):e1003481. doi: 10.1371/journal.pmed.1003481. eCollection 2021 Jan. PMID 33428616
- [Background] Garland, E. L., Kiken, L. G., Faurot, K., Palsson, O., & Gaylord, S. A. (2017). Upward spirals of mindfulness and reappraisal: Testing the mindfulness-to-meaning theory with autoregressive latent trajectory modeling. Cognitive Therapy and Research, 41(3), 381-392. https://doi.org/10.1007/s10608-016-9768-y
- [Background] Goldberg SB, Tucker RP, Greene PA, Davidson RJ, Wampold BE, Kearney DJ, Simpson TL. Mindfulness-based interventions for psychiatric disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2018 Feb;59:52-60. doi: 10.1016/j.cpr.2017.10.011. Epub 2017 Nov 8. PMID 29126747
- [Background] Hirshberg MJ, Goldberg SB, Rosenkranz M, Davidson RJ. Prevalence of harm in mindfulness-based stress reduction. Psychol Med. 2022 Apr;52(6):1080-1088. doi: 10.1017/S0033291720002834. Epub 2020 Aug 18. PMID 32807249
- [Background] Kaliman P. Epigenetics and meditation. Curr Opin Psychol. 2019 Aug;28:76-80. doi: 10.1016/j.copsyc.2018.11.010. Epub 2018 Nov 22. PMID 30522005
- [Background] Kaliman P, Alvarez-Lopez MJ, Cosin-Tomas M, Rosenkranz MA, Lutz A, Davidson RJ. Rapid changes in histone deacetylases and inflammatory gene expression in expert meditators. Psychoneuroendocrinology. 2014 Feb;40:96-107. doi: 10.1016/j.psyneuen.2013.11.004. Epub 2013 Nov 15. PMID 24485481
- [Background] Khoury B, Knauper B, Schlosser M, Carriere K, Chiesa A. Effectiveness of traditional meditation retreats: A systematic review and meta-analysis. J Psychosom Res. 2017 Jan;92:16-25. doi: 10.1016/j.jpsychores.2016.11.006. Epub 2016 Nov 18. PMID 27998508
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Kring, A. M., & Sloan, D. M. (2009). Mindfulness and emotion regulation. Emotion regulation and psychopathology: A transdiagnostic approach to etiology and treatment: Guilford Press.
- [Background] Lindsay EK, Young S, Smyth JM, Brown KW, Creswell JD. Acceptance lowers stress reactivity: Dismantling mindfulness training in a randomized controlled trial. Psychoneuroendocrinology. 2018 Jan;87:63-73. doi: 10.1016/j.psyneuen.2017.09.015. Epub 2017 Oct 8. PMID 29040891
- [Background] Lomas T, Ivtzan I, Fu CH. A systematic review of the neurophysiology of mindfulness on EEG oscillations. Neurosci Biobehav Rev. 2015 Oct;57:401-10. doi: 10.1016/j.neubiorev.2015.09.018. Epub 2015 Oct 9. PMID 26441373
- [Background] Lutz J, Herwig U, Opialla S, Hittmeyer A, Jancke L, Rufer M, Grosse Holtforth M, Bruhl AB. Mindfulness and emotion regulation--an fMRI study. Soc Cogn Affect Neurosci. 2014 Jun;9(6):776-85. doi: 10.1093/scan/nst043. Epub 2013 Apr 5. PMID 23563850
- [Background] Magan D, Yadav RK. Psychoneuroimmunology of Meditation. Ann Neurosci. 2022 Apr;29(2-3):170-176. doi: 10.1177/09727531221109117. Epub 2022 Jul 11. PMID 36419515
- [Background] Malinowski P. Neural mechanisms of attentional control in mindfulness meditation. Front Neurosci. 2013 Feb 4;7:8. doi: 10.3389/fnins.2013.00008. eCollection 2013. PMID 23382709
- [Background] Morton, M. L., Helminen, E. C., & Felver, J. C. (2020). A Systematic Review of Mindfulness Interventions on Psychophysiological Responses to Acute Stress. Mindfulness, 11(9), 2039-2054. https://doi.org/10.1007/s12671-020-01386-7
- [Background] Ostafin, B. D., Robinson, M. D., & Meier, B. P. (Eds.). (2015). Handbook of mindfulness and self-regulation. New York: Springer.
- [Background] Roca P, Vazquez C, Diez G, Brito-Pons G, McNally RJ. Not all types of meditation are the same: Mediators of change in mindfulness and compassion meditation interventions. J Affect Disord. 2021 Mar 15;283:354-362. doi: 10.1016/j.jad.2021.01.070. Epub 2021 Feb 2. PMID 33578349
- [Background] Tang YY, Holzel BK, Posner MI. The neuroscience of mindfulness meditation. Nat Rev Neurosci. 2015 Apr;16(4):213-25. doi: 10.1038/nrn3916. Epub 2015 Mar 18. PMID 25783612
- [Background] Venditti S, Verdone L, Reale A, Vetriani V, Caserta M, Zampieri M. Molecules of Silence: Effects of Meditation on Gene Expression and Epigenetics. Front Psychol. 2020 Aug 11;11:1767. doi: 10.3389/fpsyg.2020.01767. eCollection 2020. PMID 32849047
- [Background] Wielgosz J, Goldberg SB, Kral TRA, Dunne JD, Davidson RJ. Mindfulness Meditation and Psychopathology. Annu Rev Clin Psychol. 2019 May 7;15:285-316. doi: 10.1146/annurev-clinpsy-021815-093423. Epub 2018 Dec 10. PMID 30525995
- [Derived] Diez GG, Martin-Subero I, Zangri RM, Kulis M, Andreu C, Blanco I, Roca P, Cuesta P, Garcia C, Garzon J, Herradon C, Riutort M, Baliyan S, Venero C, Vazquez C. Epigenetic, psychological, and EEG changes after a 1-week retreat based on mindfulness and compassion for stress reduction in healthy adults: Study protocol of a cross-over randomized controlled trial. PLoS One. 2023 Nov 17;18(11):e0283169. doi: 10.1371/journal.pone.0283169. eCollection 2023. PMID 37976257